CLINICAL TRIAL: NCT06300281
Title: Comparison of Neuromuscular and Aquatic Exercise Programs on Fall Risk and Physical Function in Geriatrics
Acronym: NE-AEinGR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alanya Alaaddin Keykubat University (Other)
Collaborators: Pamukkale University (Other)
Responsible Party: Principal Investigator, Ozum Cetinkaya, PT, MSC. ,Principal Investigator, Alanya Alaaddin Keykubat University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NEAEGeriatircs
Record Dates: First submitted 2024-02-26; First posted 2024-03-08 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Geriatrics; Exercise Therapy; Fall; Physical Functional Performance
Keywords: Geriatrics; Exercise Therapy; Fall; Physical Functional Performance
MeSH Terms: interventions — Muscle Stretching Exercises; Aquatic Therapy

STUDY DESIGN:
Intervention Model Description: The study will be divided into two parallel groups: The neuromuscular exercise group and the Aquatic exercise group. Both groups will participate in exercise programs for 12 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Exercise Group (Experimental): A 12-week Neuromuscular exercise program consisting of sensorimotor system training, postural stability and control, global and local joint stabilization, balance training, muscle strength, breathing, and functional movement patterns will be created for the participants in Group 1.
  Interventions: Behavioral: Neuromuscular Exercise
- Aquatic Exercise Group (Experimental): Group 2 will undergo a 12-week aquatic exercise program at Alanya Alaaddin Keykubat University in a 140 cm deep pool and 32-degree water temperature.
  Interventions: Behavioral: Aquatic Exercise

INTERVENTIONS:
Behavioral: Neuromuscular Exercise — A Neuromuscular exercise program consisting of sensorimotor system training, postural stability and control, global and local joint stabilization
  Arms: Neuromuscular Exercise Group
Behavioral: Aquatic Exercise — The exercise program will begin with a 10-minute warm-up period, including straight, sideways, back walking, cycling without equipment on the parallel bar, lower extremity strength exercises, standing on tiptoes and pressing on the heels, weight transfer, resistant exercises with auxiliary devices, calisthenic exercises, hamstring and quadriceps femoris stretching. It will end with a cooling period including exercises.
  Other Names: Aquatherapy; Aquatic Rehabilitation
  Arms: Aquatic Exercise Group

SUMMARY:
Objective: The aim of this study is to compare neuromuscular and aquatic Exercise programs on fall risk and physical function in geriatrics.

Methods: As a result of the power analysis (G-Power), 36 participants are planned to be included in this study Block randomization will be used to divide participants into 2 groups, each with at least 18 participants: Group 1 (NE Group) and Group 2 (AE Group) (Randomizer.org). NE (Neuromuscular Exercise) group will participate in a 12-week exercise program consisting of sensorimotor system training, postural stability and control, global and local joint stabilization, balance training, muscle strength, breathing, and functional movement patterns.AE (Aqıuatic Exercise) Group will participate in an aquatic exercise program, which includes warm-up, mobility and strength, stretching, and cooling exercises in a 140 cm deep pool with a water temperature of 32 °. Data will be collected using the International Physical Activity Survey Short Form (IPAQ-SF), Montreal Cognitive Assessment Scale (MoCA), Geriatric Pain Measure, Optojump-next (Microgate, Bolzano, Italy), 6-minute Walk Test, 30-second-Sit-to-Stand Test, Four Step Square Test, Berg Balance Scale, Fear of Falling Avoidance Behavior Questionnaire.

Practice Implications: This current study will contribute to the understanding of how neuromuscular exercises affect falls and physical function in geriatrics.

DETAILED DESCRIPTION:
Human aging is a complex and individual process that occurs in biological, psychological, and social areas. The metabolic and physicochemical characteristics of cells gradually change with age, a process known as biological aging. This results in cellular self-regulation, regeneration, and structural alterations as well as the degeneration of healthy tissues and organs.

Physical performance impairments are linked to a wide range of negative health consequences, including osteoporosis, falls, and fractures, and are one of the most important health problems in geriatrics. Proprioceptive perception is significantly related to postural stability. Musculoskeletal system disorders (in physiological, neurological, kinesthetic, auditory, vestibular proprioception, and cognitive systems) cause balance problems, which may lead to an increase in the frequency of falls in the elderly. Exercise is critical for healthy aging and may improve walking and balance and reduce the risk of falls in the geriatric population.

Neuromuscular exercise is a relatively broad class of exercise programs that include programs aimed at improving balance, muscle activation, functional alignment, and functional joint stability, known by terms such as functional exercise, proprioceptive, agility, or perturbation training. Unlike traditional strength training, neuromuscular exercise addresses the quality of movement and emphasizes joint control in all three planes. The primary goal of neuromuscular exercise is to achieve compensatory functional stability and improve sensorimotor control. Neuromuscular exercises have been researched in knee osteoarthritis and patellofemoral pain, anterior cruciate ligament injury, fibromyalgia, obesity, autism spectrum disorder in children, cancer, chronic pain, and in various sports fields to improve balance and physical performance after injury.

Aquatic exercises are mostly rehabilitation-oriented practices that can be applied at different temperatures and depths, structured according to a specific goal. In aquatic exercises, the buoyancy of the water reduces the load on the joints, and thanks to the hydrostatic pressure providing support and resistance, older adults can exercise with a lower risk of injury and pain. Studies have shown the positive effects of aquatic exercises on improving dynamic balance, reducing the risk of falling, lower extremity strength, and mental-physical health in geriatrics.

In the literature review on the subject, no study was found comparing neuromuscular exercise and aquatic exercises in the field of geriatrics.

The aim of this study is to compare neuromuscular and aquatic Exercise programs on fall risk and physical function in geriatrics.

Methods:

Participants:

Volunteer individuals who met the inclusion and exclusion criteria and are first and second-year students of Alanya Alaaddin Keykubat University 60+ Renewal University will participate in the study. Detailed information about the study will be given to each participant who wishes to participate in the study, and their written and verbal consent will be obtained.

According to the power analysis made with the G-power program, it was found that 80% power can be obtained with 95% confidence when at least 30 people are included in the study. While calculating the sample size, timed get-up and walk test results [Group 1: 7.81 (standard deviation: 0.91), Group 2: 9.31 (standard deviation: 1.24)] were taken as a basis and the effect size was calculated as = 1.379. The risk of case loss was taken into account by taking a reserve rate of 20%, and it was planned to include 36 participants. The cases will be divided into 2 groups by block randomization using the internet program, consisting of at least 18 individuals: Group 1 [NE group] and Group 2 [AE group] (Randomizer.org).

Study Protocol:

The study will be divided into two parallel groups: The neuromuscular exercise group and the Aquatic exercise group. Both groups will participate in exercise programs for 12 weeks.

Evaluations will be administered before and after exercise programs. Data will be collected using the International Physical Activity Survey Short Form (IPAQ-SF), Montreal Cognitive Assessment Scale (MoCA), Geriatric Pain Measure, Optojump-next (Microgate, Bolzano, Italy), 6-minute Walk Test, 30-second-Sit-to-Stand Test, Four Step Square Test, Berg Balance Scale, Fear of Falling Avoidance Behavior Questionnaire.

Training and Exercise Applications:

A Neuromuscular exercise program consisting of sensorimotor system training, postural stability and control, global and local joint stabilization, balance training, muscle strength, breathing, and functional movement patterns will be created for the participants in Group 1. Exercises will start with breathing and a 10-minute warm-up period, static and dynamic proprioception, kinesthesia training (weighting on the extremities, balance, walking, open kinetic chain, closed kinetic chain exercises), postural control exercises, Frenkel coordination exercises, balance exercises (balance ball). and with a balance board), muscle strength (calisthenic exercises, therabat exercises), plyometric exercises, and core stabilization exercises will be applied progressively over the weeks and will end with a 10-minute cooling period including flexibility and relaxation exercises.

Participants in Group 2 will undergo an aquatic exercise program at Alanya Alaaddin Keykubat University in a 140 cm deep pool and 32-degree water temperature. The exercise program will begin with a 10-minute warm-up period, including straight, sideways, back walking, cycling without equipment on the parallel bar, lower extremity strength exercises, standing on tiptoes and pressing on the heels, weight transfer, resistant exercises with auxiliary devices, calisthenic exercises, hamstring and quadriceps femoris stretching. It will end with a cooling period including exercises.

Exercise sessions in both groups will last 45-60 minutes and will be applied twice a week for 12 weeks. Blood pressure measurements of all participants will be taken before the exercises. Exercise participation will be tracked in each session.

Statistical Analysis:

In the statistical analysis of data will obtain in this study, a Windows-based SPSS (IBM SPSS Statistics, Version 24.0, Armonk, NY, USA) package program will use. Continuous variables will express as a mean ± standard deviation or as a median (minimum-maximum values), and categorical variables as a number and percent. Analytical (Kolmogorov-Smirnov/Shapiro-Wilks test) and visual (Histogram and probability graphs) methods will use to test the conformity of data for normal distribution. When the parametric test assumptions were provided, Independent Sample T-Test will use to compare independent group differences; when the parametric test assumptions were not provided, the Mann Whitney-U test will use to compare independent group differences. In the dependent group analyses; when the parametric test assumptions were provided, Paired Sample T-Test will use; when the parametric test assumptions were not provided, Wilcoxon Test will use. Chi-Square Analysis and Fisher Exact Test will use compare differences between categorical variables.

ELIGIBILITY:
Inclusion Criteria:

* Being able to speak and understand Turkish,
* Getting a score at least 21 points on the Montreal Cognitive Assessment Scale (MoCA),
* Being able to walk without using any assistive device,
* Being able to adapt to the training program and wanting to participate in the study voluntarily

Exclusion Criteria:

* Presence of neurological, musculoskeletal, inner ear or eye diseases that will cause functional disability and impaired standing balance,
* Those who have had changes in their medical treatments in the last 6 months,
* Those with a history of lower extremity surgery as it may affect balance tests,
* Volunteers who do not attend at least one of the training and evaluations for any reason.
* Volunteers who want to leave the study voluntarily.
* Volunteers who cannot continue working due to any additional disease that develops.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Change in Pain | Before exercise programs and immediately after 12 weeks.
  Change in Pain will be evaluated using Geriatric Pain Measure.Geriatric Pain Scale consists of 24 items. Scores range from 0-100, scores less than 0-30 indicate mild pain; Moderate pain between 30-69 points; A score of 70 points and above is considered severe pain.
Change in walking and reaction time | Before exercise programs and immediately after 12 weeks.
  Change in walking and reaction time will be evaluated using Optojump-next (Microgate, Bolzano, Italy)
Change in aerobic capacity | Before exercise programs and immediately after 12 weeks.
  Change in aerobic capacity will be evaluated using 6-minute Walk Test
Change in muscular fitness | Before exercise programs and immediately after 12 weeks.
  Change in muscular fitness will be evaluated using 30-second-Sit-to-Stand Test
Change in s balance | Before exercise programs and immediately after 12 weeks.
  Change in static balance will be evaluated using Berg Balance Scale
Change in dynamic balance | Before exercise programs and immediately after 12 weeks.
  Change in static and dynamic balance will be evaluated using Four Step Square Test
Change in fear of falling | Before exercise programs and immediately after 12 weeks.
  Change in fear of falling will be evaluated using Fear of Falling Avoidance Behavior Questionnaire. The scale consists of thirty items and ten sub-dimensions. Sub-scores and the total score are calculated by dividing the given score by the number of items on the scale scored according to a 4-point Likert scoring. A high score indicates a high risk of falling.

SECONDARY OUTCOMES:
Physical activity level | before 12-week exercise programs
  Physical activity level will be evaluated using International Physical Activity Survey Short Form (IPAQ-SF). As a result of the test, metabolic equivalent (met) is calculated. High met indicates high physical activity.
Level of cognition | before 12-week exercise programs
  Level of cognition will be evaluated using Montreal Cognitive Assessment Scale (MoCA). Scale scores range from 0-30. A score of 21 points and above indicates a normal level of cognition.

CONTACTS AND LOCATIONS:
Overall Officials: Özüm ÇETİNKAYA, PT, MSc, Principal Investigator — Alanya Alaaddin Keykubat University; Ummuhan BAŞ ASLAN, Prof.Dr.PT., Study Director — Pamukkale University; Özgür NALBANT, Asst.Prof.Dr, Study Chair — Alanya Alaaddin Keykubat Univercity
Locations (1):
- Alanya Alaaddin Keykubat University, Alanya, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silva NC, Silva MC, Guimaraes MG, Nascimento MBO, Felicio LR. Effects of neuromuscular training and strengthening of trunk and lower limbs muscles in women with Patellofemoral Pain: A protocol of randomized controlled clinical trial, blinded. Trials. 2019 Oct 11;20(1):586. doi: 10.1186/s13063-019-3650-7. PMID 31604478
- [Background] Ageberg E, Roos EM. Neuromuscular exercise as treatment of degenerative knee disease. Exerc Sport Sci Rev. 2015 Jan;43(1):14-22. doi: 10.1249/JES.0000000000000030. PMID 25390299
- [Background] Shariat A, Ghayour Najafabadi M, Ghannadi S, Nakhostin-Ansari A, Hakakzadeh A, Shaw BS, Ingle L, Cleland JA. Effects of aquatic therapy on balance in older adults: a systematic review and meta-analysis. Eur Geriatr Med. 2022 Apr;13(2):381-393. doi: 10.1007/s41999-021-00577-2. Epub 2021 Nov 24. PMID 34817841
- [Background] Dziechciaz M, Filip R. Biological psychological and social determinants of old age: bio-psycho-social aspects of human aging. Ann Agric Environ Med. 2014;21(4):835-8. doi: 10.5604/12321966.1129943. PMID 25528930
- [Background] Pavasini R, Guralnik J, Brown JC, di Bari M, Cesari M, Landi F, Vaes B, Legrand D, Verghese J, Wang C, Stenholm S, Ferrucci L, Lai JC, Bartes AA, Espaulella J, Ferrer M, Lim JY, Ensrud KE, Cawthon P, Turusheva A, Frolova E, Rolland Y, Lauwers V, Corsonello A, Kirk GD, Ferrari R, Volpato S, Campo G. Short Physical Performance Battery and all-cause mortality: systematic review and meta-analysis. BMC Med. 2016 Dec 22;14(1):215. doi: 10.1186/s12916-016-0763-7. PMID 28003033
- [Background] Lee A, Lee KW, Khang P. Preventing falls in the geriatric population. Perm J. 2013 Fall;17(4):37-9. doi: 10.7812/TPP/12-119. No abstract available. PMID 24361019
- [Background] Scarneo SE, Root HJ, Martinez JC, Denegar C, Casa DJ, Mazerolle SM, Dann CL, Aerni GA, DiStefano LJ. Landing Technique Improvements After an Aquatic-Based Neuromuscular Training Program in Physically Active Women. J Sport Rehabil. 2017 Jan;26(1):8-14. doi: 10.1123/jsr.2015-0052. Epub 2016 Aug 24. PMID 27632861